CLINICAL TRIAL: NCT02692677
Title: An Open-Label Phase 1 Study to Determine the Absorption, Metabolism, and Routes of Excretion Following Oral Administration of (14C) Radiolabeled JNJ-42756493 to Healthy Male Subjects
Brief Title: A Study to Assess the Absorption, Metabolism, and Routes of Excretion Following Oral Administration of (14C) Radiolabeled JNJ--42756493 to Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR108125; 42756493EDI1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42756493
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- JNJ-42756493 (Experimental): Each participant will receive a single oral dose of 12 milligram (mg) of unlabeled JNJ-42756493 admixed with 14C JNJ-42756493 at Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Interventions: Drug: JNJ-42756493

INTERVENTIONS:
Drug: JNJ-42756493 — Participants will receive a single oral solution at a dose of 12 milligram (mg) of unlabeled JNJ--42756493 admixed with 14C- labeled JNJ--42756493.

SUMMARY:
The purpose of this study is to assess the absorption, metabolism, and excretion of JNJ-42756493 in healthy male adult participants after administration of a single oral dose of 12 milligram (mg) of unlabeled JNJ-42756493 admixed with 14C JNJ-42756493.

DETAILED DESCRIPTION:
This is a single--center, open--label (The researchers and participants know the treatment the participant is receiving) study. The study consists of 3 parts: Screening (35 days ), Open-label Treatment Phase (Day 1 up to Day 14 or 28); and Follow-up (up to 30 days). Total duration of the study is approximately 79 to 93 days. Plasma and urine will be collected for determination of JNJ-42756493 concentrations. Participants will be primarily evaluated for absorption, the metabolic pathways and the excretion of JNJ-42756493. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to adhere to the prohibitions and restrictions specified in the protocol
* A man who is sexually active must agree to use a condom; and a man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use a condom in combination with an adequate contraception method as deemed appropriate by the investigator (example, double-barrier method, partner using effective contraception [defined as hormonal contraception (pill, patch, injection), intrauterine device, surgical sterilization] and to not donate sperm for 5 months after receiving the study drug
* Body mass index (BMI; weight [kg]/height2 [m]2) between 18 and 30 kilogram per square meter (kg/m2) (inclusive), and body weight not less than 50 kg

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency [creatinine clearance below 90 milliliter per minute (mL/min)], thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History or current evidence of ophthalmic disorder, such as central serous retinopathy or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) and clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at screening or at admission to the study center as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 14 days before dosing is scheduled until End-of-Study procedures
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) (DSM-IV) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and Day -2 of the treatment period.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Apparent Clearance (CL/F) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vd/F) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vd/F) is influenced by the fraction absorbed.
Elimination Rate Constant | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Unbound Maximum Observed Plasma Concentration (Cmax) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The Cmax is the maximum observed plasma concentration.
Unbound Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Amount of Drug Excreted in Urine (Ae) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The Ae is the amount of drug excreted in urine. It is calculated by multiplying the urinary volume with the urinary drug concentration.
Renal Clearance (CLR) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Renal clearance calculated as Ae/AUC (last).
Area Under First Moment Plasma Concentration-Time Curve (AUMC) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  AUMC is defined as the area under first moment plasma concentration-time curve from time of dosing up to definite time t, to infinity, or to the time of last measurable concentration determined by the following equation: AUMC(0 to infinity)=Cntn/k elimination(el) + Cn/k(el^2) summation[(tn - tn^-1) (Cn^-1) (tn^-1)] + Cntn/2 where Cn=last quantifiable concentration, tn=time at which Cn is measured, k=rate constant.
Elimination Half-Life Associated With the Terminal Slope | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve, calculated as 0.693/Lamda(z).
Percentage of Drug Excreted in Urine (Ae%dose) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  The Ae%dose is the percentage of drug dose excreted into the urine calculated as (Ae divided by dose)∗100.
Amount of Drug Excreted in Urine (Ae) from t1 to t2 | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Amount of drug excreted into urine over a given time interval from t1 to t2, where t1 and t2 are the start and end times of the interval.
Percentage of Extrapolated Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (Percentage AUCinfinity, extrapolated [%AUCinf,ex]) | Pre-dose,0.5,1,2,3,4,8,12 hour post-dose(pd) on Day 1;24,36 h pd on Day 2;48 h pd on Day 3,72 h pd on Day 4; 96 h pd on Day 5;192 h pd on Day 9,216 h pd on Day 10,240 h pd on Day 11,264 h pd on Day 12,288 h pd on Day 13 and 312 h pd on Day 14
  Percentage of the AUCinfinity obtained by extrapolation calculated by ratio between AUCinfinity minus AUClast versus AUCinfinity.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Baseline up to follow up (79 to 93 days)
  An adverse event AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Madison, Wisconsin, United States